CLINICAL TRIAL: NCT00607646
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Question 3
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 Diabetes Mellitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HP-00044672-DHEA; R01DK069803-03 (NIH)
Record Dates: First submitted 2008-01-16; First posted 2008-02-06 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes
Keywords: hypoglycemia; dehydroepiandrosterone
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Hyperinsulinemic (high dose insulin) hypoglycemic clamp studies with oral administration of DHEA or placebo prior to each clamp x 2 on day 1. Day 2 hyperinsulinemic hypoglycemia. Participant randomized to either DHEA or placebo for baseline trial (arm 1) and 6 weeks treatment.
  Interventions: Drug: Dehydroepiandrosterone
- 2 (Experimental): Following 6 weeks randomized treatment, Day 1 hyperinsulinemic hypoglycemic clamps x 2 with DHEA or placebo dose given prior to each clamp. Day 2 hypoglycemia with prior dose of randomized treatment.
  Interventions: Drug: Dehydroepiandrosterone
- Arm 3 (optional) (Experimental): Individuals will be asked to return after at least 2 months and repeat the trial they did not complete (for example, placebo if they were in the DHEA trial before). Again Day 1 would consist of two hyperinsulinemic clamps with placebo or DHEA given orally. Day 2 hyperinsulinemic hypoglycemic clamp with oral administration of placebo or DHEA.
  Interventions: Drug: Placebo
- Arm 4 (Experimental): Following 6 weeks randomized treatment, Day 1 hyperinsulinemic hypoglycemic clamps x 2 with DHEA or placebo dose given prior to each clamp. Day 2 hypoglycemia with prior dose of randomized treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dehydroepiandrosterone — Placebo tablets or tablets containing DHEA will be given orally before each hyperinsulinemic clamps on day 1 (x 2). Placebo tablets or tablets containing DHEA will be given orally before Day 2 hyperinsulinemic hypoglycemic clamp x 1.
  Other Names: DHEA
  Arms: 1; 2
Drug: Placebo — Placebo oral administration prior to each clamp period x2 on day 1. Hyperinsulinemic hypoglycemia on day 2.
  Arms: Arm 3 (optional); Arm 4

SUMMARY:
Elevations of plasma cortisol, a stress hormone, during prior episodes of low blood sugar (hypoglycemia) appear to be responsible for the deficient responses during subsequent hypoglycemia. Our specific aim is to determine if dehydroepiandrosterone (DHEA), a hormone with anti-corticosteroid actions, can prevent hypoglycemia associated autonomic failure in type 1 diabetic volunteers.

DETAILED DESCRIPTION:
DHEA is the acronym for dehydroepiandrosterone, a steroid hormone produced naturally from cholesterol in the adrenal glands of males and females. It is also sold as an over-the-counter dietary supplement, and seems to have anticorticosteroid effects. DHEA antagonizes the effects of corticosterone on hippocampal function in rats and reduces responses to neural stress in mice. In our lab we have found that administration of the DHEA to rats during antecedent hypoglycemia, preserves counter-regulatory responses to subsequent hypoglycemia. The purpose of this study is to determine if the same response occurs in humans.

ELIGIBILITY:
Inclusion Criteria:

* 28 (14 males, 14 females) Healthy volunteers aged 18-45 yr.
* 28 (14 males, 14 females) Type 1 diabetic patients aged 18-45 yr.
* HbA1c < 11.0%
* Has been diagnosed Type 1 DM
* No major diabetic tissue complications (i.e. history of retinopathy, neuropathy, stasis ulcers, etc)
* Body mass index < 40kg/m-2

Exclusion Criteria:

- pregnancy

Medical history-

* Hepatic Failure/Jaundice
* Renal Failure
* Acute Cerebrovascular/ Neurological deficit

Physical Exam-

* Pneumonia
* Fever greater than 38.0 C
* Blood labs according to protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Change in level of catecholamines in blood from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States